CLINICAL TRIAL: NCT02749513
Title: Feasibility of Itraconazole as a Targeted Therapy for Inhibition of Hedgehog Pathway Signaling in Patients With Esophageal Cancer
Brief Title: Itraconazole as a Targeted Therapy for Inhibiting Hedgehog Pathway Signaling in Esophageal Cancer Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dallas VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Wang, Staff Physician, Hematology-Oncology, Dallas VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15-084
Record Dates: First submitted 2016-04-14; First posted 2016-04-25 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Itraconazole (Experimental): Itraconazole 300 mg po bid for 14-17 days
  Interventions: Drug: Itraconazole

INTERVENTIONS:
Drug: Itraconazole

SUMMARY:
The purpose of this study is to demonstrate that orally administered itraconazole, a commonly used antifungal medication, can inhibit Hedgehog pathway signaling in patients with esophageal cancer, including adenocarcinoma (EAC) and squamous cell carcinoma (ESCC).

ELIGIBILITY:
Inclusion Criteria:

• Clinical diagnosis of esophageal cancer, including gastroesophageal junction cancer

Exclusion Criteria:

* Patients unwilling or unable to provide informed consent
* Coagulopathy that precludes safe endoscopic/surgical procedure (platelet count <100,000/mm3, INR>1.5)
* Esophageal varices
* Comorbidity (e.g. pulmonary, cardiac, renal, or liver disease) that precludes safe participation in the study
* QTc>450 ms
* LFT's>3xULN
* Pregnancy
* Allergy to itraconazole
* History of symptomatic congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-01; Primary Completion 2019-09 (Actual); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Inhibition of Hedgehog pathway signaling as measured by real-time PCR. | 2-3 weeks
  mRNA expression levels as measured by real-time PCR of Hedgehog pathway ligands and target genes will be compared between baseline and post-itraconazole treatment.

SECONDARY OUTCOMES:
Inhibition of VEGFR2 pathway signaling as measured by Western blot | 2-3 weeks
  Protein expression levels of phosphorylated VEGFR2 will be compared between baseline and post-itraconazole treatment.

CONTACTS AND LOCATIONS:
Overall Officials: David Wang, MD, PhD, Principal Investigator — North Texas Veterans Healthcare System
Locations (1):
- Dallas VA Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kim DJ, Kim J, Spaunhurst K, Montoya J, Khodosh R, Chandra K, Fu T, Gilliam A, Molgo M, Beachy PA, Tang JY. Open-label, exploratory phase II trial of oral itraconazole for the treatment of basal cell carcinoma. J Clin Oncol. 2014 Mar 10;32(8):745-51. doi: 10.1200/JCO.2013.49.9525. Epub 2014 Feb 3. PMID 24493717
- [Result] Antonarakis ES, Heath EI, Smith DC, Rathkopf D, Blackford AL, Danila DC, King S, Frost A, Ajiboye AS, Zhao M, Mendonca J, Kachhap SK, Rudek MA, Carducci MA. Repurposing itraconazole as a treatment for advanced prostate cancer: a noncomparative randomized phase II trial in men with metastatic castration-resistant prostate cancer. Oncologist. 2013;18(2):163-73. doi: 10.1634/theoncologist.2012-314. Epub 2013 Jan 22. PMID 23340005
- [Derived] Zhang W, Bhagwath AS, Ramzan Z, Williams TA, Subramaniyan I, Edpuganti V, Kallem RR, Dunbar KB, Ding P, Gong K, Geurkink SA, Beg MS, Kim J, Zhang Q, Habib AA, Choi SH, Lapsiwala R, Bhagwath G, Dowell JE, Melton SD, Jie C, Putnam WC, Pham TH, Wang DH. Itraconazole Exerts Its Antitumor Effect in Esophageal Cancer By Suppressing the HER2/AKT Signaling Pathway. Mol Cancer Ther. 2021 Oct;20(10):1904-1915. doi: 10.1158/1535-7163.MCT-20-0638. Epub 2021 Aug 10. PMID 34376577